CLINICAL TRIAL: NCT02602197
Title: The Efficacy of Intravenous Paracetamol Versus Dexketoprofen for Postoperative Pain Management After Septoplasty: A Prospective Randomized Double Blind Study
Brief Title: Intravenous Paracetamol Compared Dexketoprofen for Postoperative Analgesia After Septoplasty
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Esra Caliskan, Associated Professor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA 13/100
Record Dates: First submitted 2015-03-31; First posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Pain
Keywords: Paracetamol; Dexketoprofen; postoperative pain; septoplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol (Active Comparator): 1 gr paracetamol received intravenously bolus 15 minutes after anesthetic induction and at the postoperative 6 th,12 th, 18 th and 24 th hours
  Interventions: Drug: Paracetamol
- Dexketoprofen (Active Comparator): 50 mg dexketoprofen received intravenous bolus 15 minutes after anesthetic induction and at the postoperative 8 th,16 th and 24 th hours.
  Interventions: Drug: Dexketoprofen

INTERVENTIONS:
Drug: Paracetamol — After anesthetic induction, the first I.V bolus injections of 1 gr paracetamol (total amount of 100 ml) were given during 15 minutes and then repeated every 6 h until 24 h postoperative period.
  Other Names: Parol
  Arms: Paracetamol
Drug: Dexketoprofen — After anesthetic induction, the first I.V bolus injections of 50 mg Dexketoprofen (premixed with 0.9 % sodium chloride to total amount of 100 ml) were given during 15 minutes and then repeated every 8 h until 24 h postoperative period.
  Other Names: Arveles
  Arms: Dexketoprofen

SUMMARY:
The investigators conducted a prospective, randomized, double blind study to compare the effectiveness of intravenous paracetamol and dexketoprofen for preventing pain during first 24 hours postoperative period in adult patient undergoing septoplasty.

DETAILED DESCRIPTION:
Postoperative pain scores as measured by Visual Analog Scale (VAS) (0 represented no pain and 10 the worst pain ever experienced) at 15, 30, 60 minutes and 2th, 4th, 6th, 12th and 24th hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* After patient's inform consent was approved, a total of 70 ASA (American Society of Anesthesiology) physical status I and II adult patients age 18 to 65 undergoing septoplasty were planned include the study.

Exclusion Criteria:

* History of clotting disorders or blood dyscrasias,
* Gastrointestinal ulcer or chronic dyspepsia,
* History of allergy to the study drugs,
* Active bleeding or bleeding disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change from pain scores until postoperative 24 hours | Pain scores recorded during postoperative 24 hours.
  Pain scores as measured by Visual Analog Scale (VAS) at 15 and 30 minutes, 1h, 2h, 4h, 6h, 12h, and 24 h after surgery

SECONDARY OUTCOMES:
Cumulative tramadol consumption during postoperative 24 hours. | First postoperative 24 hours
  Cumulative tramadol consumption was recorded during postoperative 24 hours.